CLINICAL TRIAL: NCT06822400
Title: A Multi-center, Randomized, Controlled Investigation of Tetralogy of Fallot in Neonates
Brief Title: Investigation of Tetralogy of Fallot in Neonates
Acronym: RIFAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Children's Hospital of Fudan University (Other); Suzhou University Affiliated Children's Hospital (Other); Shenzhen Children's Hospital (Other Government); West China Second University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20241226
Record Dates: First submitted 2025-01-02; First posted 2025-02-12 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Tetralogy of Fallot (TOF); Pulmonary Stenosis; Ventricular Septal Defects (VSD); Double Outlet Right Ventricle
Keywords: Neonatal; Infant; RCT; surgery
MeSH Terms: conditions — Tetralogy of Fallot; Pulmonary Valve Stenosis; Heart Septal Defects, Ventricular; Double Outlet Right Ventricle | interventions — Parturition; Aging

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator)
  Interventions: Procedure: corrective surgery within 28 days of birth
- control group (Placebo Comparator)
  Interventions: Procedure: corrective surgery between 3-6 months of age

INTERVENTIONS:
Procedure: corrective surgery within 28 days of birth — Participants will be randomized into two groups with a 1:1 allocation:
  Intervention Group: Neonates undergoing surgical correction of TOF within 28 days of birth.
  Arms: intervention group
Procedure: corrective surgery between 3-6 months of age — Participants will be randomized into two groups with a 1:1 allocation:
  Control Group: Infants undergoing surgical correction of TOF between 3-6 months of age
  Arms: control group

SUMMARY:
Child health serves as the foundation for overall public health, with neonatal mortality recognized globally as a comprehensive indicator of national health standards and societal advancement. The Healthy Children Action Improvement Plan (2021-2025) sets a national target to reduce neonatal mortality in China to below 3.1‰. Congenital heart disease (CHD), the most prevalent congenital defect among neonates, constitutes a significant cause of disability and premature death in the Chinese population. Annually, approximately 70,000-80,000 neonates are born with CHD, among whom nearly 10,000 present with critical congenital heart disease (CCHD). Postnatal manifestations of CCHD often include cyanosis, hypoperfusion, and respiratory distress, with untreated cases resulting in approximately 50% mortality. CCHD is one of the leading causes of infant death.

Tetralogy of Fallot (TOF), the most common form of CCHD, accounts for a substantial proportion of cyanotic congenital heart diseases. It is characterized by four anatomical abnormalities: ventricular septal defect, pulmonary stenosis, overriding aorta, and right ventricular hypertrophy. These structural defects disrupt intracardiac blood flow, reduce arterial oxygen saturation, and result in cyanosis and other related symptoms. Untreated TOF leads to significant health issues early in life, including growth retardation, recurrent hypoxic episodes, heart failure, and increased susceptibility to infections. Long-term survival is markedly reduced, with only a small proportion surviving into adulthood. Thus, surgical intervention is pivotal for improving outcomes in TOF(Tetralogy of Fallot) patients.

Despite advances in medical technology yielding satisfactory early outcomes, long-term prognosis following TOF correction remains a challenge. Historically, surgical strategies emphasized complete relief of right ventricular outflow tract obstruction, often at the expense of pulmonary valve function. Recent studies, however, highlight the critical role of preserving pulmonary valve function in improving long-term outcomes, as pulmonary valve dysfunction is a leading cause of late right ventricular failure and reintervention. Additionally, surgical approaches, whether via atrial or ventricular access, have inherent advantages and limitations, but neither can fully eliminate the risk of postoperative arrhythmias associated with TOF's anatomical complexity and surgical impact. These issues underscore the necessity for further advancements in long-term management strategies.

Surgical correction of TOF in a single-stage procedure has become standard practice, with the timing of surgery progressively shifting to earlier ages-from school age in the 1990s to the current standard of 3-6 months of age. This timing ensures sufficient weight and organ maturity to withstand the complexities of cardiac surgery. However, in clinical practice, significant challenges persist, including: (1) Deterioration during the waiting period, during which patients may experience recurrent hypoxic episodes, inadequate weight gain, and exacerbated pulmonary vascular underdevelopment, thereby complicating definitive surgery and increasing perioperative risk. (2) Developmental delays due to chronic hypoxemia and heart failure, potentially leading to neurological deficits and pulmonary hypertension, adversely affecting cognitive and motor development. Neonatal repair, performed within 28 days of life, may mitigate these challenges by restoring normal circulatory physiology at the earliest possible stage.

International guidelines endorse neonatal TOF repair for capable centers, citing the potential for enhanced clinical benefits and superior prognoses. Clinical observations at our center indicate several advantages of neonatal TOF repair, including reduced intraoperative bleeding, cleaner surgical fields, and better pulmonary vascular development. These benefits may be attributed to the regenerative potential of neonatal myocardial cells and the absence of prolonged pathological circulatory states, which otherwise exacerbate anatomical abnormalities. Early intervention may reduce right ventricular fibrosis and pulmonary vascular pathology, thereby improving long-term outcomes.

With advancements in surgical techniques and perioperative care, neonatal TOF repair has become a routine practice at our center, with over 100 cases performed annually for two consecutive years. This success is supported by an integrated prenatal-to-postnatal care model, establishing a comprehensive treatment framework.

Given this context, the investigators propose a multicenter, randomized controlled trial (RCT) to compare the safety and efficacy of neonatal and infant TOF repair. This study aims to provide high-quality evidence for clinical practice, determine optimal surgical timing, and enhance overall survival rates and quality of life for TOF patients.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of TOF's Disease. Full-term neonates aged ≤28 days. Birth weight of all eligible male or female patients >2.5 kg. All included study participants must be able to give an informed consent

Exclusion Criteria:

Preterm infants . Coexisting complex cardiac anomalies. Severe TOF with pulmonary artery hypoplasia , recurrent hypoxic episodes , or conditions warranting palliative or single-ventricle repair.

Extra-cardiac anomalies, including genetic or chromosomal abnormalities. Neonatal bronchopulmonary dysplasia. Deteriorating conditions in the control group precluding surgery by 3 months of age.

Parental refusal to participate in the clinical trial.

Ages: 1 Minute to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events(mortality) | up to 30 days
  All-cause mortality within 30 days postoperatively, encompassing cardiovascular and non-cardiovascular causes.
Rate of re-intervention 12 months after surgery | up to 12 months
  Reoperation rate within 12 months postoperatively based on defined criteria, excluding in-hospital reinterventions.

SECONDARY OUTCOMES:
Perioperative situation | during surgery
  Perioperative indicators：surgery duration in minutes
Perioperative situation | during surgery
  Perioperative indicators：bypass time in minutes
Perioperative situation | up to 720 hours
  Perioperative indicators：intensive care unit length of stay in hours
Perioperative situation | up to 720 hours
  Perioperative indicators：duration of ventilation in hours
Perioperative situation | up to 30 days
  Perioperative indicators：hospital length of stay in days
Surgical complications | up to 720 hours
  Surgical complications:postoperative ECMO support in hours
Surgical complications | up to 720 hours
  Surgical complications:peritoneal dialysis in hours
Cardiac related examination indicators | through study completion, an average of 3 year
  Echocardiographic parameter：right ventricular wall thickness in millimeters
Cardiac related examination indicators | through study completion, an average of 3 year
  Echocardiographic parameter：right ventricular outflow tract gradients in mmHg
Cardiac related examination indicators | through study completion, an average of 3 year
  Echocardiographic paramete：pulmonary regurgitation area in cm^2
Cardiac related examination indicators | through study completion, an average of 3 year
  Echocardiographic parameter：tricuspid regurgitation area in cm^2
Follow up indicators | through study completion, an average of 3 year
  weight in kilograms
Follow up indicators | through study completion, an average of 3 year
  height in meters
Follow up indicators | through study completion, an average of 3 year
  weight and height will be combined to report BMI in kg/m^2
Economic indicators | up to 30 days
  hospitalization costs in yuan
Economic indicators | during surgery
  operation costs in yuan
Economic indicators | through study completion, an average of 3 year
  medical costs in yuan during perioperative and postoperative follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes